CLINICAL TRIAL: NCT00598351
Title: A Prospective Natural History Study of Patients With Neurofibromatosis Type 2 (NF2).
Brief Title: Natural History Study of Patients With Neurofibromatosis Type 2
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080044; 08-N-0044
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-09-03

CONDITIONS: Neurofibromatosis
Keywords: Meningioma; Ependymoma; Schwannoma; Spinal Cord Tumor; Vestibular Schwannoma; Natural History
MeSH Terms: conditions — Neurofibromatoses; Meningioma; Ependymoma; Neurilemmoma; Spinal Cord Neoplasms; Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients must have the diagnosis of NF2 by established clinical criteria or genetic testing.

SUMMARY:
Objective

With this prospective natural experiment trial on neurofibromatosis type 2 (NF2) study, we hope to understand the factors leading to tumor progression and neurological disease burden in NF2.

Study Population

A total of 269 participants, ages 8-75, with a clinical or genetic diagnosis of NF2 will participate in this study.

Design

Study participants will be evaluated with a thorough physical and neurologic examination upon enrollment. This initial outpatient evaluation will include magnetic resonance imaging with contrast of brain and spine and blood collection for research use. Participants with measurable hearing will have audiology assessment performed. Participants with untreated vestibular schwannomas will have vestibular assessment performed during the initial visit. Genetic studies performed outside will be acceptable as confirmation of NF2 in enrolled patients. If needed to confirm NF2 with genetic studies, or for research purpose, whole genome/whole exome sequencing may be performed on blood obtained from subjects enrolled in this study. All participants will be evaluated by a speech language pathologist.

Subjects will be followed as outpatients for up to ten years, during which clinical, and radiologic evaluation will be performed annually. Auditory testing will be performed annually for participants with measurable hearing. Participants with initially untreated vestibular schwannomas will be followed annually with vestibular testing. Speech and swallowing reassessments will be repeated if worsening of speech or swallowing is reported. Blood will be collected at each visit for blood biomarker testing

Outcome measures

We hope to understand the biologic basis for speech and swallowing dysfunction in patients with NF2. We will study and report the strength of association of MRI findings, clinical assessments cranial nerve deficits and speech/swallowing dysfunction. We hope to

identify imaging biomarkers of hearing loss in NF2. We will attempt to discover the mode of peripheral neuropathy in patients with NF2. Lastly, we will attempt to discover previously unknown serum biomarkers associated with high tumor burden in NF2.

DETAILED DESCRIPTION:
Objective

With this prospective natural history study on neurofibromatosis type 2 (NF2) study, we hope to understand the factors leading to tumor progression and neurological disease burden in NF2.

Study Population

A total of 269 participants, ages 8-75, with a clinical or genetic diagnosis of NF2 will participate in this study.

Design

Study participants will be evaluated with a thorough physical and neurologic examination upon enrollment. This initial outpatient evaluation will include magnetic resonance imaging with contrast of brain and spine and blood collection for research use. Participants with measurable hearing will have audiology assessment performed during the initial visit. Participants with untreated vestibular schwannomas will have vestibular assessment performed during the initial visit. Genetic studies performed outside will be acceptable as confirmation of NF2 in enrolled patients. If needed to confirm NF2 with genetic studies, or for research purpose, whole genome/whole exome sequencing may be performed on blood obtained from subjects enrolled in this study. All participants will be evaluated by a speech language pathologist.

Subjects will be followed as outpatients for up to ten years, during which clinical, and radiologic evaluation will be performed annually. Auditory testing will be performed annually for participants with measurable hearing. Participants with initially untreated vestibular schwannomas will be followed annually with vestibular testing. Speech and swallowing reassessments will be repeated if worsening of speech or swallowing is reported. Blood will be collected at each visit for blood biomarker testing

Outcome measures

We hope to understand the biologic basis for speech and swallowing dysfunction in patients with NF2. We will study and report the strength of association of MRI findings, clinical assessments cranial nerve deficits and speech/swallowing dysfunction. We hope to

identify imaging biomarkers of hearing loss in NF2. We will attempt to discover the mode of peripheral neuropathy in patients with NF2. Lastly, we will attempt to discover previously unknown serum biomarkers associated with high tumor burden in NF2.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must meet all the following criteria:

* Have the diagnosis of NF2 by established clinical criteria or genetic testing.
* Be between the age of 8 and 75.
* Have the capacity to undergo serial MRI scanning of the CNS without IV sedation.
* Able to give informed consent, or have a parent able to provide informed consent if a child.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

* Have a clinically unstable condition that precludes serial clinical and imaging evaluation (i.e. Class 3 congestive heart failure, severe chronic renal insufficiency, severe chronic obstructive pulmonary disease).
* Cannot have an MRI scan due to an allergy or relative contraindication to MRI contrast agents, prior surgery or implant that involves metal clips or wires, which might be expected to cause tissue damage or produce image artifacts such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, and artificial heart valves.
* ABIs or cochlear implants are not approved by the NIH Radiology department for safe use on NIH scanners..
* Have severe chronic renal insufficiency (glomerular filtration rate less than 30 mL/min/1.73 m2), hepatorenal syndrome or post-liver transplantation.
* Are pregnant at time of intake visit (women of childbearing age will be tested with a urine pregnancy test).

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects with a diagnosis of NF2 by established clinical criteria or genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2008-03-21 (Actual)

PRIMARY OUTCOMES:
To determine the natural history (clinical and radiographic) of nervous system tumors in NF2 | annual for up to 10 years
  Clinical Variables (longitudinal: measured annually for each subject)a. Subjective speech and swallowing dysfunction (binary)b. Spinal cord function:Modified ASIA Motor Scalec. Ambulatory status:modified McCormick grading scaled. Overall function:Karnofsky Performance Statuse. NFTI-QOLf. Functional Independence Measure scale MRI Variables (longitudinal: measured annually for each subject):a. Tumor volume (continuous variable) for VS tumors, meningiomas, other schwannomas, ependymomas, and Total tumor burden (number and volume). Specific growth rates of tumors.b. FLAIR hyper-intensity MRI Variables (cross-sectional: measured at baseline and as needed for each subject):c. MRI of Right Upper and Lower Extremity Laboratory testing variables (longitudinal:measured annually for each subject):a. Audiometry Laboratory testing variables (cross-sectional:measured at baseline and as needed for each subject)b. EMG/NCV study valuesc. Vestibular testing Covariate variable:a. Ageb. Sex

SECONDARY OUTCOMES:
To identify the underlying causes, and patterns of progression of speech and swallowing problems in patients with NF2 | Annual for up to 10 years
  Self-reported swallowing deficits (binary, yes vs no) based on the last Visit (cross-sectional data)
To identify imaging biomarkers of hearing loss in patients with NF2 | Annual for up to 10 years
  MRI Variables (longitudinal: measured annually for each subject):a. Tumor volume (continuous variable) for VS tumors, meningiomas, other schwannomas, ependymomas, and Total tumor burden(number and volume). Specific growth rates of tumors.b. FLAIR hyper-intensity MRI Variables (crosssectional: measured at baseline and as needed for each subject
To identify the etiology of peripheral neuropathy in patients with NF2 | Annual for up to 10 years
  MRI images of the Right upper extremity will be evaluated for the presence of peripheral nerve lesions at baseline. These imaging findings will be evaluated with respect to EMG/NCV results.
To identify serum biomarkers of NF2 disease progression | Annual for up to 10 years
  determination of serum biomarker status and suspected biologic markers of disease progression using quantitative immunoassay or newer proteomic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-N-0044.html